CLINICAL TRIAL: NCT03200691
Title: Phase II Study of Neoadjuvant Anti-PD-1 Antibody SHR-1210 and Radiation in Resectable Esophageal Squamous Cell Carcinoma
Brief Title: Neoadjuvant Anti-PD-1 Antibody SHR-1210 and Radiation in Resectable Esophageal Squamous Cell Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hangzhou Cancer Hospital (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Shixiu Wu, Professor, Hangzhou Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HangzhouCH09
Record Dates: First submitted 2017-06-22; First posted 2017-06-27 (Actual); Last update posted 2017-08-07 (Actual); Status verified 2017-08

CONDITIONS: Esophageal Neoplasms; Esophageal Diseases
Keywords: Esophageal Squamous Cell Carcinoma; PD-1; Neoadjuvant treatment
MeSH Terms: conditions — Esophageal Neoplasms; Esophageal Diseases; Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nimotuzumab with radiotherapy (Experimental): Patients will receive neoadjuvant radiotherapy with concurrent anti-PD-1 antibody SHR-1210. Radiation of primary tumor and local lymph nodes with 95% planning target volume (PTV) of 40Gy/20f.
  SHR-1210 200mg fixed dose every 2 weeks delivered concurrent with radiation therapy.
  After 2-4 weeks of neoadjuvant treatment, patients will be evaluated by a multidisciplinary teams (MDTs) and esophagectomy will be given for patients with resectable disease.
  Interventions: Radiation: 3-DCRT or IMRT radiation; Drug: anti-PD-1 antibody SHR-1210

INTERVENTIONS:
Radiation: 3-DCRT or IMRT radiation — Radiation of primary tumor and local lymph nodes with 95% planning target volume (PTV) of 40 Gy/20f.
Drug: anti-PD-1 antibody SHR-1210 — SHR-1210 (200mg fixed dose every 2 weeks for 2 cycles) will be administered as an intravenous infusion over 60 minutes.

SUMMARY:
The objective of this study is to evaluate the efficacy and safety of radiation therapy combined with anti-PD-1 antibody SHR-1210 followed by surgery in treating patients with resectable esophageal squamous cell carcinoma

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically confirmed esophageal squamous cell carcinoma without prior treatments including surgery, chemotherapy, radiotherapy, and targeting treatment.
2. With resectable disease of primary tumor in middle or lower thoracic esophagus and clinical stage Ⅱa-Ⅲ.
3. age:18-75 years, male or female.
4. Can provide either a newly obtained or archival tumor tissue sample.
5. ECOG 0-1.
6. Life expectancy of greater than 12 weeks.
7. Without serious system dysfunction and could tolerate radiotherapy.
8. Patients must have normal marrow function with a hemoglobin (HGB) of ≥90g/L, an white blood cell (WBC) counts of ≥4.0×109/L，a neutrophil count of ≥2.0×109/L, , a platelet count of ≥100×109/L, a total bilirubin (TBil) of ≤1.5 upper normal limitation (UNL), a creatinine (Cr) of ≤ 1.5 UNL, alanine aminotransferase (ALAT) and aspartate aminotransferase (ASAT) of ≤2.5 UNL.
9. Patients must have normal electrocardiogram results and no history of congestive heart failure.
10. Women of childbearing age should voluntarily take contraceptive measures.
11. Without drug addition
12. Patients must be with good compliance and agree to accept follow-up of disease progression and adverse events
13. Patients must give written informed consent signed voluntarily by patients themselves or their supervisors witted by doctors.

Exclusion Criteria:

1. Patients who have or are currently undergoing additional chemotherapy, radiation therapy, targeted therapy or immunotherapy.
2. With unresectable disease including any T4b or M1 disease
3. Complete obstruction of the esophagus, or patients who have the potential to develop perforation
4. Other malignancy within 5 years prior to entry into the study, expect for curatively treated basal cell and squamous cell carcinoma of the skin and/or curatively resected in-situ cervical and/or breast cancers.
5. Known central nervous system (CNS) metastases.
6. Subjects with any active autoimmune disease or history of autoimmune disease.
7. Uncontrolled clinically significant heart disease, including but not limited to the following: (1) > NYHA II congestive heart failure; (2) unstable angina, (3) myocardial infarction within the past 1 year; (4) clinically significant supraventricular arrhythmia or ventricular arrhythmia requirement for treatment or intervention;
8. Active infection or an unexplained fever > 38.5°C during screening or before the first scheduled day of dosing (subjects with tumor fever may be enrolled at the discretion of the investigator);
9. History of Interstitial Pneumonia or active non-infectious pneumonitis.
10. Known Human Immunodeficiency Virus (HIV) infection、active Hepatitis B or Hepatitis C.
11. Prior therapy with a PD-1, anti-PD-Ligand 1 (PD-L1) agent.
12. Known history of hypersensitivity to macromolecular protein preparation or any components of the SHR-1210 formulation.
13. Concurrent medical condition requiring the use of cortisol (>10mg/day Prednisone or equivalent dose) or other systematic immunosuppressive medications within 14 days before the study treatment. Except: inhalation or topical corticosteroids. Doses > 10 mg/day prednisone orequivalent for replacement therapy.
14. Received a live vaccine within 4 weeks of the first dose of study medication.
15. Pregnancy or breast feeding.
16. Decision of unsuitableness by principal investigator or physician-in-charge.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2017-08-10 (Estimated); Primary Completion 2018-06-30 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
Pathologic Complete Response Rate | 2-4 weeks after completion of radiotherapy
  the Percentage of Patients Who Have No Evidence of Cancer in Their Surgical Specimen Following Surgery

SECONDARY OUTCOMES:
Disease-Free Survival | 2 years
  Defined as the interval between the start date of treatment and the date of occurrence of progressive disease or death from any cause.
Numbers of adverse events and the degree of each adverse events according to the NCI CTCAE 4.0 criteria. | 6 months
  From the date of randomization to 6 months after esophagectomy. An expected average of 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hangzhou Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No